CLINICAL TRIAL: NCT01615068
Title: An Observational Cohort Study of Treatment Patterns and Outcomes in Patients With HER2 Positive (HER2+) Metastatic Breast Cancer (SystHERs Registry (Systemic Therapies for HER2+ Metastatic Breast Cancer Study)).
Brief Title: An Observational Study in Patients With HER2 Positive Metastatic Breast Cancer (SystHERs Registry)
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28257
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and whole blood samples

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, prospective observational study will evaluate the treatment patterns, and the safety in patients with HER2-positive (HER2+) metastatic breast cancer (MBC). Eligible patients will have an initial metastatic breast cancer diagnosis that has not been previously treated with systemic therapy; patients may be enrolled up to 6 months after the diagnosis. Data will be collected for up to 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Initial diagnosis of HER2+ MBC, as diagnosed by the treating physician, no more than 6 months prior to study enrollment
* Availability of cancer-specific historical data points in the patient's medical records

Exclusion Criteria:

* Any inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2 positive (HER2+) metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2012-06-05 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Distribution of patients receiving unique treatment regimen/sequence of treatment regimens | Up to 8 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 8 years
Overall survival (OS) | Up to 8 years
Post-progression survival (PPS) | Up to 8 years
Time-to-treatment failure (TTF) | Up to 8 years
Response rate (RR) | Up to 8 years
Safety: Incidence of adverse events | Up to 8 years
Patient-reported outcome assessment (PRO) | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (142):
- United States (142):
  - St. Vincent'S Hospital; Birmingham Hematology Oncology Associates, Llc, Birmingham, Alabama
  - University of South Alabama; Mitchell Cancer Institute, Mobile, Alabama
  - Arizona Oncology Associates, PC - NAHOA, Sedona, Arizona
  - Arizona Oncology, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - East Valley Hem/Onc Med Group; Metropolitan Hem Onc., Burbank, California
  - South Bay Oncology Hematology Partners, Campbell, California
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - ROBERT A. MOSS, M.D., F.A.C.P., Inc, Fountain Valley, California
  - California Oncology of the Central Valley, Fresno, California
  - Cancer Care Associates, Fresno, California
  - St. Jude Heritage Healthcare; Virgiia K.Crosson Can Ctr, Fullerton, California
  - University of Southern California, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Comprehensive Cancer Care, Palm Springs, California
  - Univ of Calif, San Francisco; Breast Cancer Center, San Francisco, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Medical Oncology, Santa Maria, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Center - Denver, Denver, Colorado
  - Mile High Oncology, Littleton, Colorado
  - Connecticut Oncology Group, Middletown, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Hematology Oncology P.C., Stamford, Connecticut
  - MedStar Washington Hosp Center, Washington D.C., District of Columbia
  - Lynn Cancer Institute - West, Boca Raton, Florida
  - University of Miami; Dept Sylvester Cancer Center, Deerfield Beach, Florida
  - Florida Cancer Specialists - Fort Myers (New Hampshire Ct), Fort Myers, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Baptist - MD Anderson Cancer Center, Jacksonville, Florida
  - Florida Oncology Associates, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Md Anderson Cancer Center Orlando, Orlando, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Florida Cancer Specialists (St. Petersburg - St. Anthony's Professional Building), St. Petersburg, Florida
  - Space Coast Medical Associates, Titusville, Florida
  - Peachtree Hematology & Oncology Consultants, Pc, Atlanta, Georgia
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Summit Cancer Care PC, Savannah, Georgia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Alton Memorial Hospital; Outpatient Clinic and Infusion Center, Alton, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Mid-Illinois Hematology, Normal, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Oncology Hematology Assoc, Evansville, Indiana
  - McFarland Clinic, Ames, Iowa
  - University of Iowa, Iowa City, Iowa
  - Mercy Medical Ctr-North Iowa ; Mercy Cancer Center, Mason City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - James Graham Brown Cancer Center, University of Louisville, Louisville, Kentucky
  - Baptist Hospital East, Louisville, Kentucky
  - Mary Bird Perkins Cancer Ctr, Baton Rouge, Louisiana
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Lafayette General Medical Center, Lafayette, Louisiana
  - Mercy Oncology / Hematology Center; Oncology, Portland, Maine
  - Western Maryland Health Sys, Cumberland, Maryland
  - Associates in Oncology/Hematology P.C., Rockville, Maryland
  - Capitol Hematology & Oncology, Silver Spring, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - Carroll County Cancer Center, Westminster, Maryland
  - Berkshire Hematology, Oncology Pc, Pittsfield, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Southdale Cancer Clinic U of M Medical Center, Fairview- Edina, Edina, Minnesota
  - Minnesota Oncology Hematology, Pa, Minneapolis, Minnesota
  - Park Nicollet Clinic Cancer Center, Saint Louis Park, Minnesota
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Research Medical Center; Pharmacy, Kansas City, Missouri
  - Christian Hospital; Outpatient Cancer and Infusion Center, St Louis, Missouri
  - St. John'S Mercy Medical Center; David C. Pratt Cancer Center, St Louis, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Southeast Nebraska Cancer Center;; Southeast Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center; Gastroenterology Section, Lebanon, New Hampshire
  - Portsmouth Regional Hospital; Hem/Onc Clinic, Portsmouth, New Hampshire
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Onc & Hematology Specialists, Denville, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology Oncology Associates; Carol G. Simon Ctr, Morristown, New Jersey
  - Luckow Pavillion, Valley Hosp; Office of Clinical Trials, Paramus, New Jersey
  - The Mary Imogene Bassett Hospi, Cooperstown, New York
  - North Shore Hem Onc Associates, East Setauket, New York
  - Queens Hospital Center, Jamaica, New York
  - Beth Israel Comprehensive Cancer Center Pharmacy, New York, New York
  - Herbert Irving Comprehensive Cancer Center; Herbert Irving Pavillion, New York, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Gaston Hematology/Oncology, Gastonia, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - First Health of the Carolinas, Pinehurst, North Carolina
  - Metro Health Medical Center, Cleveland, Ohio
  - Mid Ohio Onc Hematology Inc, Columbus, Ohio
  - Signal Point Clinical; Research Center, LLC, Middletown, Ohio
  - Flower Memorial Hospital, Sylvania, Ohio
  - Mercy Clinic Oklahoma Communties, Inc, Oklahoma City, Oklahoma
  - Cancer Care Assoc-15th St, Tulsa, Oklahoma
  - Providence Cancer Center, Portland, Oregon
  - Hematology & Oncology Assoc; North Eastern Pennsylvania, Dunmore, Pennsylvania
  - Lancaster Cancer Center, Ltd., Lancaster, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital; Transplantation Services, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Sch of Med; Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Guthrie Clinic, Sayre, Pennsylvania
  - Charleston Hematology Oncology, Charleston, South Carolina
  - Medical Univ of South Carolina, Charleston, South Carolina
  - South Carolina Oncology Associates - SCRI, Columbia, South Carolina
  - Chattanooga Oncology and Hematology Associates, PC, Chattanooga, Tennessee
  - Kingsport Hematology Oncology Associates, Kingsport, Tennessee
  - Center for Biomedical Research LLC, Knoxville, Tennessee
  - Boston Baskin Cancer Foundation, Nashville, Tennessee
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Hendrick Cancer Center, Abilene, Texas
  - Texas Oncology, Bedford, Texas
  - St. Joseph Regional Cancer Ct, Bryan, Texas
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - Texas Oncology- El Paso Cancer Treatment Center Gateway, El Paso, Texas
  - Texas Oncology, P.A. - Fort Worth, Fort Worth, Texas
  - Texas Oncology - Houston (Gessner), Houston, Texas
  - Texas Oncology, P.A. - McAllen; South Texas Cancer Center-McAllen, McAllen, Texas
  - Texas Oncology - Paris, Paris, Texas
  - Tyler Hematololgy Oncology, PA, Tyler, Texas
  - Texas Oncology, PA, Waco, Texas
  - Texas Oncology, P.A.; Duke Slayton Cancer Center, Webster, Texas
  - Northern Utah Associates, Ogden, Utah
  - Huntsman Cancer Institute; Oncology, Salt Lake City, Utah
  - Lynchburg Hem Onc Clinic Inc, Lynchburg, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Shenandoah Oncology Associates, Winchester, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Columbia Saint Mary's; Medical Oncology, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Tripathy D, Brufsky A, Cobleigh M, Jahanzeb M, Kaufman PA, Mason G, O'Shaughnessy J, Rugo HS, Swain SM, Yardley DA, Chu L, Li H, Antao V, Hurvitz SA. De Novo Versus Recurrent HER2-Positive Metastatic Breast Cancer: Patient Characteristics, Treatment, and Survival from the SystHERs Registry. Oncologist. 2020 Feb;25(2):e214-e222. doi: 10.1634/theoncologist.2019-0446. Epub 2019 Oct 14. PMID 32043771
- [Derived] Cobleigh M, Yardley DA, Brufsky AM, Rugo HS, Swain SM, Kaufman PA, Tripathy D, Hurvitz SA, O'Shaughnessy J, Mason G, Antao V, Li H, Chu L, Jahanzeb M. Baseline Characteristics, Treatment Patterns, and Outcomes in Patients with HER2-Positive Metastatic Breast Cancer by Hormone Receptor Status from SystHERs. Clin Cancer Res. 2020 Mar 1;26(5):1105-1113. doi: 10.1158/1078-0432.CCR-19-2350. Epub 2019 Nov 26. PMID 31772121
- [Derived] Hurvitz SA, O'Shaughnessy J, Mason G, Yardley DA, Jahanzeb M, Brufsky A, Rugo HS, Swain SM, Kaufman PA, Tripathy D, Chu L, Li H, Antao V, Cobleigh M. Central Nervous System Metastasis in Patients with HER2-Positive Metastatic Breast Cancer: Patient Characteristics, Treatment, and Survival from SystHERs. Clin Cancer Res. 2019 Apr 15;25(8):2433-2441. doi: 10.1158/1078-0432.CCR-18-2366. Epub 2018 Dec 28. PMID 30593513
- [Derived] Tripathy D, Rugo HS, Kaufman PA, Swain S, O'Shaughnessy J, Jahanzeb M, Mason G, Beattie M, Yoo B, Lai C, Masaquel A, Hurvitz S. The SystHERs registry: an observational cohort study of treatment patterns and outcomes in patients with human epidermal growth factor receptor 2-positive metastatic breast cancer. BMC Cancer. 2014 May 2;14:307. doi: 10.1186/1471-2407-14-307. PMID 24885258